CLINICAL TRIAL: NCT00366717
Title: Cytomegalovirus Reactivation in Cancer Patients Receiving Chemotherapy
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Other Study IDs: MMH-I-S-144
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2006-08-21 (Estimated); Status verified 2006-01

CONDITIONS: Cancer; Cytomegalovirus
Keywords: Cancer under chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Cytomegalovirus (CMV) infects most of the world population. This study is to understand if chemotherapy will increase the chance of reactivating CMV. The results may help us in determining when treatment is needed and perhaps Why is it needed.

DETAILED DESCRIPTION:
Despite CMV reactivation has been clearly described in patients underwent transplantation, this phenomenon has not been studied in patients undergoing chemotherapy. Our purpose is to understand if CMV number increases in monocytic leukocytes during chemotherapy and how is the host response to that changes.

Virus load will be studied by quantitative PCR, host response will be studied by measuring patient's anti-CMV IgG, CMV-associated symptoms, serum IFN-r and TNF-a.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of any cancer
* chemotherapy is needed for more than 6 months
* age>20 years old

Exclusion Criteria:

* those who do not agree to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-06; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ta Lu, MD, PhD., Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- See also: Home page of Mackay Memorial Hospital — http://www.mmh.org.tw